CLINICAL TRIAL: NCT03364543
Title: The UTHealth Medical-Legal Partnership: Improving Health by Addressing Health-Harming Legal Needs
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Winston Liaw, Associate Professor, The University of Texas Health Science Center, Houston
Other Study IDs: 2017-048
Record Dates: First submitted 2017-11-30; First posted 2017-12-06 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Social Determinants of Health

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Medical-Legal Partnership Group: The Medical-Legal Partnership Group are lawyers in clinics who address health-harming legal needs. This group will also have access to access to a social worker and a community worker.
  Interventions: Other: Access to the Medical-Legal Partnership Group; Other: Access to social worker and a community worker
- Usual Care: Access to a social worker and a community worker, but no systematic process for addressing health-harming legal needs.
  Interventions: Other: Access to social worker and a community worker

INTERVENTIONS:
Other: Access to the Medical-Legal Partnership Group — The Medical-Legal Partnership Group are lawyers in clinics who address health-harming legal needs.
  Groups: Medical-Legal Partnership Group
Other: Access to social worker and a community worker — Access to social worker and a community worker, but no systematic process for addressing health-harming legal needs.

SUMMARY:
The purpose of this study is to assess the acceptability, feasibility, and preliminary effectiveness of the UTHealth medical-legal partnerships (MLP) against usual care.

ELIGIBILITY:
Inclusion Criteria:

* English- or Spanish- speaking
* screen positive for health-harming legal needs (HHLNs)

Exclusion Criteria:

* Those unable or unwilling to consent to legal services

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: These are adults patients accessing primary care clinics.
Sampling Method: Non-Probability Sample
Enrollment: 911 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Number of participants who had an emergency department visit | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Winston Liaw, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (2):
- United States (2):
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - UTHealth Comprehensive Sickle Cell Center, Houston, Texas